CLINICAL TRIAL: NCT06130345
Title: Post-marketing Safety of Elasomeran/Davesomeran and Andusomeran Vaccines in the United States
Brief Title: Post-marketing Safety of Elasomeran/Davesomeran and Andusomeran
Status: Completed | Type: Observational
Sponsor: ModernaTX, Inc. (Industry)
Collaborators: Aetion, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: mRNA-1273-P920
Record Dates: First submitted 2023-11-08; First posted 2023-11-14 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: SARS-CoV-2
Keywords: Elasomeran; Davesomeran; Andusomeran; SARS-CoV-2; SARS-CoV-2 Vaccine; Coronavirus; Virus Diseases; Messenger RNA; COVID-19; COVID-19 Vaccine; Moderna
MeSH Terms: conditions — Coronavirus Infections; Virus Diseases; COVID-19 | interventions — 2019-nCoV Vaccine mRNA-1273; CVnCoV COVID-19 vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort 1: Influenza Vaccinated Concurrent Comparator: Participants who receive an elasomeran/davesomeran or an andusomeran vaccine in routine clinical practice are compared to participants who receive an influenza vaccine to observe differences in the rate of adverse events of special interest during an etiologically relevant window.
  Interventions: Biological: SPIKEVAX
- Cohort 2: Medically Attended COVID-19 Concurrent Comparator: Participants who receive an elasomeran/davesomeran or an andusomeran vaccine in routine clinical practice are compared to participants who diagnosed with COVID-19 to observe differences in in the rate of adverse events of special interest during an etiologically relevant window.
  Interventions: Biological: SPIKEVAX

INTERVENTIONS:
Biological: SPIKEVAX — Intramuscular injection
  Other Names: SARS-CoV-2-mRNA vaccine; SPIKEVAX Bivalent; Spikevax XBB.1.5; Elasomeran; Davesomeran; Andusomeran

SUMMARY:
The main objective of the study is to evaluate the safety of the elasomeran/davesomeran and andusomeran vaccines as used in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1: Influenza vaccinated concurrent comparator

Eligible vaccine episodes must meet the following inclusion criteria within the protocol-specified time windows:

* Non-missing sex: (start of available data, 1 day prior to index)
* No receipt of elasomeran/davesomeran and andusomeran vaccine: (90 days prior to index, 1 day prior to index)
* No receipt of influenza vaccine: (90 days prior to index, 1 day prior to index)
* No receipt of any other COVID-19 vaccine: (90 days prior to index, index date)
* Continuous enrollment in closed medical and pharmacy claims (365 days prior to index, index date)

Cohort 2: Medically attended COVID-19 concurrent comparator

Eligible vaccine and disease episodes must meet the following inclusion criteria within the specified time windows:

* Non-missing sex: (start of available data, 1 day prior to index)
* No receipt of elasomeran/davesomeran and andusomeran vaccine: (180 days prior to index, 1 day prior to index)
* No evidence of medically attended COVID-19: (180 days prior to index, 1 day prior to index)
* No receipt of any other COVID-19 vaccine: (180 days prior to index, index date)
* Continuous enrollment in closed medical and pharmacy claims (365 days prior to index, index date)

Exclusion Criteria:

* Vaccine and disease episodes with a prior AESI within the washout window will be excluded from the analytic cohort.
* For the influenza vaccinated concurrent comparator cohort, individuals who receive an elasomeran/davesomeran and andusomeran vaccine and an influenza vaccine on the same day or within a minimum number of days will be excluded from the primary analysis.

Note: Other protocol-defined inclusion/exclusion criteria may apply.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be identified using HealthVerity's aggregated medical and pharmacy claims database between September 1, 2022 and February 29, 2024.
Sampling Method: Non-Probability Sample
Enrollment: 15196685 (Actual)
Dates: Start 2023-04-14 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events of Special Interest (AESI) | Day 2 up to Day 60 after vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Aetion, Inc, New York, New York, United States